CLINICAL TRIAL: NCT04346862
Title: Phase IV Study to Evaluate the Effect of Improvement in Cognitive Impairment of Acetyl-L-carnitine in Patients With Mild Cognitive Impairment Accompanied With Chronic Cerebrovascular Disease
Brief Title: Evaluation the Effect of Acetyl-L-carnitine in Patients With Mild Cognitive Impairment Accompanied With Chronic Cerebrovascular Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM-VASCA-401
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetyl-L-carnitine hydrochloride (Experimental)
  Interventions: Drug: Acetyl-L-carnitine hydrochloride 500mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetyl-L-carnitine hydrochloride 500mg — The participants will receive treatment of Acetyl-L-carnitine hydrochloride 500mg, orally, 3 times a day for 24weeks
  Arms: Acetyl-L-carnitine hydrochloride
Drug: Placebo — The participants will receive treatment of placebo of Acetyl-L-carnitine hydrochloride 500mg, orally, 3 times a day for 24weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of Acetyl-L-carnitine in patient with Mild Cognitive Impairment associated with chronic cerebrovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Age between 55 and 85 years old
* Patients with chronic cerebrovascular disease, who have modified Fazekas scale grade 2 ~ 3
* Patients wtih a diagnosis of MCI
* MOCA-K of 23 or less
* Patients who provided a signed written informed consent form

Exclusion Criteria:

* Patiens who are uneducated or illiterate
* Patiens previously treated with dementia
* Patients who received a nootropic agent or thyroid hormone within 4 weeks of visit 1
* Patients with cognitive impairment due to diseases other than cerebrovascular disease
* Patients with severe depression, schizophrenia, alcoholism, and drug dependence

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Estimated)
Dates: Start 2016-01-26 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Interference score using K-CWST(Korean-Color Word Stroop Test) | 24 week
  interference score is defined as 'the time required to test stage 2(Color-Word)' minus ''the time required to test stage 1(Word)
Montreal Cognitive Assessment Korean(MOCA-K) | 24 week
  MOCA-K included cognitive domains; attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. MOCA-K scored from 0 to 30. The higher the score, the better.

SECONDARY OUTCOMES:
Korean Trail Making Test Elderly(K-TMT-e) | 24 week
  The K-TMT-e was composed of 2 parts: part A calls for the test-taker to connect randomly distributed numbers (1-25) on a test paper in ascending order (1->2->3...), whereas part B requires the test-taker to alternate numbers and letters (1->A->2->B...).
EQ-5D | 24 week
  EQ-5D included 5 dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Clinical Global Impression -Improvement (CGI-I) | 24 week
  CGI-I scored from 1 (very much improved) to 7 (very much worse).

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic Kwandong University International St. Mary'S Hospital, Incheon, South Korea